CLINICAL TRIAL: NCT02590120
Title: Comparaison du Profil d'Absorption Des Acides aminés Entre Une Nutrition entérale Semi-élémentaire et Une Nutrition entérale polymérique
Brief Title: Enteral Nutrition and Amino Acid Absorption
Acronym: PEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 12.02.FR.NHS
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-03

CONDITIONS: Malabsorption
MeSH Terms: conditions — Malabsorption Syndromes | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enteral nutrition product : product A (Active Comparator): Administration during 16 hours.
  Interventions: Dietary Supplement: Enteral nutrition
- Enteral nutrition product : product B (Active Comparator): Administration during 16 hours.
  Interventions: Dietary Supplement: Enteral nutrition

INTERVENTIONS:
Dietary Supplement: Enteral nutrition

SUMMARY:
The purpose of this study is to evaluate amino acid absorption with two different type of proteins.

ELIGIBILITY:
Inclusion Criteria:

* Patient with gastrointestinal disorder : citrulline plasma concentration < 20 µmol/L and/or xylose plasma concentration < 1,7 mmol/L
* Patient under enteral nutrition at home
* Patient already receiving 1 L by day

Exclusion Criteria:

* Obese patient BMI > 30
* Diabetes
* Renal or liver failure
* Glucocorticoids treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Amino acid absorption profile | 48 hours
  Area under the curve of amino acid plasma concentration

SECONDARY OUTCOMES:
Tolerance | 48 hours
  Description and occurence of adverse events
Nutritional status | 48 hours
  Retinol Binding Protein and Transthyretin dosage
Essentials amino acid absorption | 48 hours
  Area under the curve of plasma concentration
Insulinemia evolution | 48 hours
  Insulinemia dosage
Link between amino acid and insuline | 48 hours
  Correlation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Julien Gautry, MD, Study Chair — Nestle Health Science
Locations (1):
- CHU de Lille, Lille, France